CLINICAL TRIAL: NCT02251990
Title: A Phase III Randomized Multinational Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172/MK-8742 in Treatment-Naïve Subjects With Chronic HCV GT 1, GT 4 and GT 6 Infection
Brief Title: Grazoprevir (MK-5172) and Elbasvir (MK-8742) Combination in Treatment-Naïve Hepatitis C Virus Participants (MK-5172-067)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-067
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment Group (ITG): Grazoprevir/Elbasvir (Experimental): Participants receive a grazoprevir/elbasvir FDC tablet once daily (q.d.) by mouth during a 12-week Active Treatment period (Week 1 to Week 12) and are followed-up for 24 weeks to Week 36.
  Interventions: Drug: Grazoprevir/Elbasvir
- Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir (Placebo Comparator): Participants receive a placebo tablet q.d. by mouth for 12 weeks (placebo treatment period). After a 4-week Follow-Up period, participants receive open-label grazoprevir/elbasvir FDC during a 12-week Active Treatment period (Week 16 to Week 28). Participants are then followed-up for 24 weeks to Week 52.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Grazoprevir/Elbasvir — FDC tablet containing 100 mg of grazoprevir and 50 mg of elbasvir taken q.d. by mouth for 12 weeks.
  Other Names: MK-5172A
  Arms: Immediate Treatment Group (ITG): Grazoprevir/Elbasvir
Drug: Placebo — Placebo tablet matching grazoprevir/elbasvir FDC tablet taken q.d. by mouth for 12 weeks.
  Arms: Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir

SUMMARY:
This is a randomized, parallel-group, placebo-controlled, multi-site, multinational, double-blind followed by open label period, Phase 3 trial of 100 mg of grazoprevir (MK-5172) in combination with 50 mg of elbasvir (MK-8742) (grazoprevir/elbasvir fixed-dose combination [FDC]) in treatment-naïve (TN) participants with chronic hepatitis C virus (HCV), genotype (GT) 1, 4 or 6 infection. The primary hypothesis is that the percentage of participants receiving grazoprevir/elbasvir FDC in the Immediate Treatment Group (ITG) achieving Sustained Virologic Response 12 weeks after the end of all study therapy (SVR12) will be superior to the historical reference rate of 73%.

ELIGIBILITY:
Inclusion Criteria:

* Has documented chronic HCV GT1, GT4, or GT6 (with no evidence of non-typeable or mixed genotype) infection
* Meets clinical criteria for presence or absence of cirrhosis based on liver disease staging assessment
* Is abstinent or uses acceptable method(s) of contraception

Exclusion Criteria:

* Has evidence of decompensated liver disease
* Is coinfected with hepatitis B virus or human immunodeficiency virus (HIV)
* Shows evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* Has a clinically-relevant drug or alcohol abuse within 12 months of screening
* Is pregnant or breast-feeding
* Has any condition or abnormality that might confound the results of the trial or pose an additional risk to the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Wei L, Jia JD, Wang FS, Niu JQ, Zhao XM, Mu S, Liang LW, Wang Z, Hwang P, Robertson MN, Ingravallo P, Asante-Appiah E, Wei B, Evans B, Hanna GJ, Talwani R, Duan ZP, Zhdanov K, Cheng PN, Tanwandee T, Nguyen VK, Heo J, Isakov V, George J; C-CORAL Investigators. Efficacy and safety of elbasvir/grazoprevir in participants with hepatitis C virus genotype 1, 4, or 6 infection from the Asia-Pacific region and Russia: Final results from the randomized C-CORAL study. J Gastroenterol Hepatol. 2019 Jan;34(1):12-21. doi: 10.1111/jgh.14509. Epub 2018 Dec 9. PMID 30311701
- [Result] George J, Burnevich E, Sheen IS, Heo J, Kinh NV, Tanwandee T, Cheng PN, Kim DY, Tak WY, Kizhlo S, Zhdanov K, Isakov V, Liang L, Lindore P, Ginanni J, Nguyen BY, Wahl J, Barr E, Robertson M, Ingravallo P, Talwani R; C-CORAL Study Investigators. Elbasvir/grazoprevir in Asia-Pacific/Russian participants with chronic hepatitis C virus genotype 1, 4, or 6 infection. Hepatol Commun. 2018 Apr 4;2(5):595-606. doi: 10.1002/hep4.1177. eCollection 2018 May. PMID 29761174
- [Derived] Dalgard O, Litwin AH, Shibolet O, Grebely J, Nahass R, Altice FL, Conway B, Gane EJ, Luetkemeyer AF, Peng CY, Iser D, Gendrano IN, Kelly MM, Haber BA, Platt H, Puenpatom A; CO-STAR Investigators. Health-related quality of life in people receiving opioid agonist treatment and treatment for hepatitis C virus infection. J Addict Dis. 2023 Jul-Sep;41(3):213-224. doi: 10.1080/10550887.2022.2088978. Epub 2022 Aug 3. PMID 35920743
- [Derived] Wei L, Jia JD, Duan ZP, Wang FS, Niu JQ, Xie W, Huang WX, Zhang MX, Huang Y, Wang MR, Wu SM, Zhao YR, Jia ZS, Zhao XM, Mu SM, Liang LW, Wang Z, Puenpatom A, Hwang P, Robertson MN, Ingravallo P, Asante-Appiah E, Wei B, Evans B, Hanna GJ, Talwani R. Efficacy and safety of elbasvir/grazoprevir in treatment-naive Chinese adults with hepatitis C virus infection: A randomized trial. JGH Open. 2020 Jul 15;4(6):1065-1073. doi: 10.1002/jgh3.12387. eCollection 2020 Dec. PMID 33319038
- [Derived] Asselah T, Reesink H, Gerstoft J, de Ledinghen V, Pockros PJ, Robertson M, Hwang P, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Talwani R, Serfaty L. Efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 4 infection: A pooled analysis. Liver Int. 2018 Sep;38(9):1583-1591. doi: 10.1111/liv.13727. Epub 2018 Mar 31. PMID 29461687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Subject Disposition, Period 1 covers Day 1 through Week 12 for both treatment groups. Period 2 covers Week 12 through Week 36 for the Immediate Treatment Group (ITG) and Week 12 through Week 28 for the Deferred Treatment Group (DTG). Period 3 covers Week 28 through Week 52 for the DTG; the ITG completed the study with Period 2.
Pre-assignment Details: A total of 489 participants were randomized to treatment, and 488 participants received ≥1 dose of study drug during the blinded period. One participant randomized to the ITG withdrew consent after randomization, but prior to receiving study drug.
Groups:
- Immediate Treatment Group (ITG): Grazoprevir/Elbasvir: Participants received a grazoprevir/elbasvir fixed-dose combination (FDC) tablet once daily (q.d.) by mouth during a 12-week Active Treatment period (Week 1 to Week 12) and were followed-up for 24 weeks to Week 36.
- Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir: Participants received a placebo tablet q.d. by mouth for 12 weeks (placebo treatment period). After a 4-week Follow-Up period, participants received open-label grazoprevir/elbasvir FDC during a 12-week Active Treatment period (Week 16 to Week 28). Participants were then followed-up for 24 weeks to Week 52.
Period: Period 1 (Double-blind [DB])
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir
Started | 366 | 123
Treated | 365 (Started Grazoprevir/Elbasvir) | 123 (Started Placebo)
Completed | 358 (Completed 12 weeks of Grazoprevir/Elbasvir) | 122 (Completed 12 weeks of Placebo)
Not Completed | 8 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not Treated | 1 | 0
Period: Period 2 (ITG Follow-up/DTG Open Label)
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir
Started | 360 (2 participants that did not complete Period 1 treatment were included in Follow-up.) | 121 (1 participant completing Period 1 was not eligible for Period 2 and was not treated.)
Completed | 360 (Completed 24 weeks of follow-up) | 118 (Completed 12 weeks of Grazoprevir/Elbasvir)
Not Completed | 0 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 0 | 2
Period: Period 3 (DTG Follow-up)
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir
Started | 0 (The ITG completed the study with Period 2) | 121 (3 participants that discontinued treatment in Period 2 were included in Follow-up.)
Completed | 0 | 121 (Completed 24 weeks of follow-up)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study treatment.
Groups:
- Immediate Treatment Group (ITG): Grazoprevir/Elbasvir: Participants received a grazoprevir/elbasvir FDC tablet q.d. by mouth during a 12-week Active Treatment period (Week 1 to Week 12) and were followed-up for 24 weeks to Week 36.
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir | Total
Number analyzed (Participants) | 365 | 123 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (12.9) | 48.6 (12.9) | 48.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 67 | 272
  Male | 160 | 56 | 216

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After the End of All Study Therapy (SVR12)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS® AmpliPrep/COBAS® Taqman HCV Test, v2.0, which had a lower limit of quantification (LLOQ) of 15 IU/mL. SVR12 was defined as HCV RNA below the lower limit of detection (<LLOQ) at 12 weeks after the end of all study therapy. As pre-specified in the protocol, the Deferred Treatment Group was not included in the primary efficacy analysis.
Time Frame: 12 weeks after end of all therapy (Study Week 24)
Population: All randomized participants in the Immediate Treatment Group who received at least one dose of study treatment. The Deferred Treatment Group was not included in the primary efficacy analysis.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 365 | 0
percentage of participants | 94.2 [91.5 to 97.0] |
Statistical Analysis 1: Comparison: Immediate Treatment Group (ITG): Grazoprevir/Elbasvir; A one-sided Wald test was used to test the null hypothesis, which was that the SVR12 rate for the ITG was ≤ the historical reference rate of 73%. The historical reference SVR rate for treatment-naive genotype 1 predominantly Asian participants treated with pegylated interferon/ribavirin was derived from 2 studies (PMCID: PMC417, PMCID: PMC3644280) after adjusting for an expected improved safety profile related to an interferon-free regimen; Test type: Superiority or Other; p < 0.001, one-sided asymptotic test — The p-value was based on a one-sided asymptotic test for a binomial proportion. A one-sided p-value <0.0125 was considered supportive of a conclusion that the true SVR12 is >73%

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event (AE) During the DB Treatment Period and First 14 Follow-up Days
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that is temporally associated with the use of the Sponsor's product, is also an AE. The primary safety analysis compared the safety data of the Immediate Treatment Group during the active treatment period to those of the Deferred Treatment Group during the placebo treatment period.
Time Frame: DB Treatment period plus first 14 follow-up days (up to 14 weeks)
Population: All randomized participants who received at least one dose of study treatment during the double-blind treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 365 | 123
percentage of participants | 50.7 | 51.2
Statistical Analysis 1: Comparison: Immediate Treatment Group (ITG): Grazoprevir/Elbasvir vs Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir; Estimates and 95% CIs were calculated for between-treatment differences (ITG minus DTG) in the percentage of participants with events using the Miettinen and Nurminen method; Test type: Superiority or Other; Difference in Percentages = -0.5, 95% CI 2-sided [-10.6 to 9.6]

3. Primary Outcome: Percentage of Participants That Discontinued From Study Therapy Due to AEs During the DB Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that is temporally associated with the use of the Sponsor's product, is also an AE. A participant could discontinue from treatment but continue to participate in the study as long as consent was not withdrawn. The primary safety analysis compared the safety data of the Immediate Treatment Group during the active treatment period to those of the Deferred Treatment Group during the placebo treatment period.
Time Frame: DB Treatment period (up to 12 weeks)
Population: All randomized participants who received at least one dose of study treatment during the double-blind treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 365 | 123
percentage of participants | 0.3 | 0.8
Statistical Analysis 1: Comparison: Immediate Treatment Group (ITG): Grazoprevir/Elbasvir vs Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Percentages = -0.5, 95% CI 2-sided [-4.2 to 0.9]

4. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After the End of All Study Therapy (SVR24)
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS® AmpliPrep/COBAS® Taqman HCV Test, v2.0, which had a LLOQ of 15 IU/mL. SVR24 was defined as HCV RNA <LLOQ at 24 weeks after the end of all study therapy. As pre-specified in the protocol, the Deferred Treatment Group was not included in the secondary efficacy analysis.
Time Frame: 24 weeks after end of all therapy (Study Week 36)
Population: All randomized participants in the Immediate Treatment Group who received at least one dose of study treatment. The Deferred Treatment Group was not included in the secondary efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 365 | 0
percentage of participants | 94.0 [91.5 to 96.4] |

5. Other Pre Specified Outcome: Percentage of Participants Achieving Sustained Virologic Response 4 Weeks After the End of All Study Therapy (SVR4)
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS® AmpliPrep/COBAS® Taqman HCV Test, v2.0, which had a LLOQ of 15 IU/mL. SVR4 was defined as HCV RNA <LLOQ at 4 weeks after the end of all study therapy. As pre-specified in the protocol, the Deferred Treatment Group was not included in this efficacy analysis.
Time Frame: 4 weeks after end of all therapy (Study Week 16)
Population: All randomized participants in the Immediate Treatment Group who received at least one dose of study treatment. The Deferred Treatment Group was not included in this efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo > Grazoprevir/Elbasvir
Number analyzed (Participants) | 365 | 0
percentage of participants | 96.2 [94.2 to 98.1] |

ADVERSE EVENTS:
Time Frame: Immediate Treatment Group = Up to Week 36; Deferred Treatment: Placebo Group = Up to Week 16; Deferred Treatment: Grazoprevir/Elbasvir Group = Week 16 to Week 52
Description: All randomized participants who received ≥1 dose of study treatment and had any safety follow-up data. AEs were reported by the treatment that participants were receiving at the time of the event; AEs for Deferred Group reported separately for placebo and active treatment periods.
Groups:
- Deferred Treatment Group (DTG): Placebo: Participants received a placebo tablet q.d. by mouth for 12 weeks during the double-blind treatment period (Weeks 1 to 12). Participants were then followed-up for 4 weeks to Week 16.
- Deferred Treatment Group (DTG): Grazoprevir/Elbasvir: Participants received open-label grazoprevir/elbasvir FDC during a 12-week Active Treatment period (Week 16 to Week 28). Participants were then followed-up for 24 weeks to Week 52.
Arm/Group | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir | Deferred Treatment Group (DTG): Placebo | Deferred Treatment Group (DTG): Grazoprevir/Elbasvir
Serious Adverse Events (participants affected / at risk) | 9/365 | 3/123 | 6/121
Other Adverse Events (participants affected / at risk) | 85/365 | 30/123 | 21/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir (N=365) | Deferred Treatment Group (DTG): Placebo (N=123) | Deferred Treatment Group (DTG): Grazoprevir/Elbasvir (N=121)
Evans syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment Group (ITG): Grazoprevir/Elbasvir (N=365) | Deferred Treatment Group (DTG): Placebo (N=123) | Deferred Treatment Group (DTG): Grazoprevir/Elbasvir (N=121)
Diarrhoea (Gastrointestinal disorders) | 21 (22) | 8 (8) | 3 (3)
Fatigue (General disorders) | 21 (21) | 8 (8) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 26 (30) | 8 (9) | 10 (10)
Alanine aminotransferase increased (Investigations) | 6 (6) | 7 (7) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 7 (9) | 4 (4)
Headache (Nervous system disorders) | 24 (24) | 6 (11) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.